CLINICAL TRIAL: NCT05194787
Title: TAS Test: Determining the Feasibility and Validity of Online Motor-cognitive Testing for Early Detection of Alzheimer's Disease
Brief Title: TAS Test: Online Motor-cognitive Tests for Early Detection of Alzheimer's Disease
Acronym: TASTest
Status: Recruiting | Type: Observational
Sponsor: University of Tasmania (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Sydney (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, Jane Alty, Associate Professor of Neurology, University of Tasmania
Other Study IDs: H0021660
Record Dates: First submitted 2021-12-29; First posted 2022-01-18 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease; Dementia; Age-related Cognitive Decline
Keywords: pre-clinical; early detection; online tests; Artificial intelligence
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for p-tau 181 and APOE4
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cognitive test scores, clinical diagnosis and blood biomarkers — Clinical diagnosis of Alzheimer's disease, mild cognitive impairment or normal ageing.
  Cognitive test score on CANTAB Blood biomarker (p-tau 181) level

SUMMARY:
Global dementia prevalence is rising. Alzheimer's disease (AD), the most common cause, has devastating effects on people's quality of life. AD has a preclinical (pre-AD) period of 10-20 years when brain pathology silently progresses before any cognitive symptoms appear. Current tests for pre-AD are invasive, costly and unsuitable for screening at population level. Similar to screening for pre-diabetes and carcinoma in situ, it is important to detect AD at the preclinical stage in order to offer early interventions before the pathology progresses to the irrerversible degenerative stage. In the study, research will develop a new scalable test (TAS Test) by combining two innovative ideas: hand-movement tests to detect pre-AD >10 years before cognitive symptoms begin; and computer vision so people can "self-test" online using home computers. This unique approach builds on recent discoveries that hand-movement patterns change in pre-AD. The research team will use exquisitely precise computer vision methods to automatically analyse movement data from thousands of participants, and combine this with machine learning of overall motor-cognitive performance. The project team has access to 3 well-phenotyped cohorts, >10,000 existing participants and a cutting-edge assay for a blood AD biomarker, ptau181. The research team will develop a TAS Test algorithm to classify hand-movement and cognitive test data for pre-AD risk (p-taua181 levels) and determine TAS Test's precision to prospectively predict 5-year risks of cognitive decline and AD.

DETAILED DESCRIPTION:
Sub-study 1: Cross-sectional study design: From two established cohorts with pre-existing datasets of up to 10 years of longitudinal cognitive, genetic and demographic data, the team will recruit 500 participants over 50 years old who are confirmed to have normal cognition. At baseline and months 3 and 6, the participants will be invited to complete TAS Test online at home, or in the research centre if preferred. The participants will also have a baseline blood test for ptau181 levels (and APOE4 if required). The research team will integrate movement data to develop a multivariable model that discriminates between pre-AD (positive p-tau181) and normal cognitive ageing (negative p-tau181).

Sub-study 2: Prospective 5-year cohort study design: The researchers will invite 10,000 adults from an established long-term (ISLAND Project) cohort to complete online tests at home: (i) TAS Test every 6 months, and (ii) Cambridge Neuropsychological Test Automated Battery (CANTAB) cognitive tests every 24 months. The prospective 'high risk' predictions of TAS Test at baseline will be validated against CANTAB scores, and also clinically (face to face gold standard consensus diagnosis of AD vs MCI vs normal) in a subsample of 300.

ELIGIBILITY:
Inclusion Criteria: > 50years old

Exclusion Criteria: established diagnosis of dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Currently focused on adults aged > 50 years in established cohort studies in Australia: ie participants from Tasmanian Healthy Brain Project, Healthy Brain and Ageing project or ISLAND Project.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Develop and validate the optimal TAS Test protocol to detect pre-AD (p-tau 181 positivity) | 3 years
  Receiver Operating Characteristic (ROC) curves will be plotted against the positive p-tau181 cut-off to assess the sensitivity/specificity of TAS Test models to identify the pre-AD stage.
Prospectively validate TAS Test to predict risks of cognitive decline | 5 years
  Assess the sensitivity and specificity of TAS Test to predict cognitive trajectories (CANTAB scores) "stable" and "declining" using ROC curve analysis.
Prospectively validate TAS Test to predict risks of AD diagnosis | 5 years
  Multinomial logistic regression will estimate the (covariate adjusted) log-odds of being in each diagnostic category (AD, MCI and normal) at 5 years as predicted by baseline TAS Test results.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Vickers, PhD DSc, Study Director — University of Tasmania; A/Prof Bai, PhD MSc, Principal Investigator — University of Tasmania
Locations (1):
- University of Tasmania, Hobart, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alty J, Bai Q, Li R, Lawler K, St George RJ, Hill E, Bindoff A, Garg S, Wang X, Huang G, Zhang K, Rudd KD, Bartlett L, Goldberg LR, Collins JM, Hinder MR, Naismith SL, Hogg DC, King AE, Vickers JC. The TAS Test project: a prospective longitudinal validation of new online motor-cognitive tests to detect preclinical Alzheimer's disease and estimate 5-year risks of cognitive decline and dementia. BMC Neurol. 2022 Jul 18;22(1):266. doi: 10.1186/s12883-022-02772-5. PMID 35850660
- See also: University profile for Principal Investigator — https://www.utas.edu.au/profiles/staff/health/jane-alty